CLINICAL TRIAL: NCT05308160
Title: A Single Center, Randomized, Open Label, Parallel Group, Phase 3 Study to Evaluate the Efficacy of Dapagliflozin in Subjects With Nonalcoholic Fatty Liver Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202104098MIPC
Record Dates: First submitted 2022-03-07; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-06

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Active Comparator): This trial is a randomized, open label, two-arm, parallel-group, non-used comparator, single center trial to evaluate the efficacy of dapagliflozin in subjects with Nonalcoholic fatty liver disease.
  Interventions: Drug: Dapagliflozin 10Mg Tab
- Non-used drug (Placebo Comparator): This trial is a randomized, open label, two-arm, parallel-group, non-used comparator, single center trial to evaluate the efficacy of dapagliflozin in subjects with Nonalcoholic fatty liver disease.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — This trial is a randomized, open label, two-arm, parallel-group, non-used comparator, single center trial to evaluate the efficacy of dapagliflozin in subjects with Nonalcoholic fatty liver disease. This is a principal investigator initiate study. This study is supported by Liver Disease Prevention & Treatment Research Foundation. Dapagliflozin will be provided free of charge by AstraZeneca.
  Arms: Dapagliflozin
Drug: Placebo — This trial is a randomized, open label, two-arm, parallel-group, non-used comparator, single center trial to evaluate the efficacy of dapagliflozin in subjects with Nonalcoholic fatty liver disease. This is a principal investigator initiate study. This study is supported by Liver Disease Prevention & Treatment Research Foundation. Dapagliflozin will be provided free of charge by AstraZeneca.
  Arms: Non-used drug

SUMMARY:
This trial is a randomized, open label, two-arm, parallel-group, non-used comparator, single center trial to evaluate the efficacy of dapagliflozin in subjects with Nonalcoholic fatty liver disease. This is a principal investigator initiate study. This study is supported by Liver Disease Prevention & Treatment Research Foundation. Dapagliflozin will be provided free of charge by AstraZeneca.

ELIGIBILITY:
Inclusion criteria

For inclusion in the study patients should fulfil the following criteria:

1. Provision of informed consent prior to the time of registration.
2. Aged 20-74 years male or female who are diagnosed with NAFLD and FibroScan shows CAP score ≥ 252 dB/m (≥Steatosis grade 2).

3.30 or more mL/min/1.73 m2 of estimated glomerular filtration rate 4.Female subjects must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception for the duration of the study (from the time they sign consent) and for 1 month after the last dose of IP to prevent pregnancy. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used.

5.Subjects who are blood donors should not donate blood during the study and for 1 month following their last dose of IP.

Exclusion criteria

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Viral hepatitis or other types of liver disorder (e.g. drug-induced or autoimmune hepatitis).
2. Alcohol consumption above recommended limits (male: more than 30g/ day; female: more than 20g/day converting to ethanol).
3. Serious liver dysfunction (Child-Pugh B or C).
4. History of any other malignancy within 1 years (with the exception of successfully treated non-melanoma skin cancers).
5. Patients with a known hypersensitivity to investigator product (IP).
6. Participation in another clinical trial within the previous 30 days or involvement in the planning and/or conduct of the study.
7. Previous enrolment or randomisation in the present study.
8. Active gallbladder diseases
9. For women is currently pregnant (confirmed with positive pregnancy test) or breast feeding.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety Outcome Measure | 6 months
  Patients who meet all inclusion criteria and none of the exclusion criteria and are not screen failures for reasons listed above will be randomized in a 1:1 ratio to either receive 10 mg per day dapagliflozin or enter control group at Visit 2.

CONTACTS AND LOCATIONS:
Locations (1):
- NTUH, Taipei, Zhongzheng Dist., Taiwan